CLINICAL TRIAL: NCT03604588
Title: Evaluation of HPV OncoTect ™ for the Etiological Diagnosis of HPV-induced Oropharyngeal Cancers
Acronym: HPV OncoTect™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01655-46; 2016/2474 (Other: CSET number)
Record Dates: First submitted 2018-07-20; First posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Oropharyngeal Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with oropharyngeal cancer (Other): Salivary specimens will be collected from 40 patients with oropharyngeal cancer The saliva samples will be sent to incell dx, which will analyze them blindly (without knowledge of the clinicopathological information) with the HPV OncoTect ™ test.
  Clinical and pathological information will be collected and maintained by the principal investigator At the end of the study, the results obtained with the HPV OncoTect ™ test will be confronted with the clinical and pathological results.
  Interventions: Diagnostic Test: HPV OncoTect™

INTERVENTIONS:
Diagnostic Test: HPV OncoTect™ — Salivary specimens will be collected from 40 patients with oropharyngeal cancer The saliva samples will be sent to incell dx, which will analyze them blindly (without knowledge of the clinicopathological information) with the HPV OncoTect ™ test.
  Clinical and pathological information will be collected and maintained by the principal investigator At the end of the study, the results obtained with the HPV OncoTect ™ test will be confronted with the clinical and pathological results.

SUMMARY:
To determine the sensitivity of HPV OncotectTM to diagnose oropharyngeal cancers induced by oncogenic HPV

ELIGIBILITY:
Inclusion Criteria:

1. Untreated oropharynx epidermoid carcinoma
2. Patient ≥ 18 years old
3. Patient affiliated to a social security scheme or beneficiary of such a scheme
4. Information to the patient or his legal representative and signature of informed consent

Exclusion Criteria:

1. Non-oropharyngeal epidermoid carcinoma
2. Oropharyngeal epidermoid carcinoma previously treated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity is defined as the probability that the oncotectTM HPV test is positive if the cancer is HPV-induced. | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No